CLINICAL TRIAL: NCT06460285
Title: CalmER Intervention Trial for Healthcare Workers With Anxiety
Brief Title: Intervention Trial for Healthcare Workers With Anxiety
Acronym: CalmER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, George M. Slavich, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#23-001651
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anxiety
Keywords: anxiety; stress; emotion regulation
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Due to the objectives and nature of the study, the identity of test and control treatments will be known to investigators and research staff. Participants will, however, be blind to their conditional assignment. The active control condition was carefully selected to ensure that participants would be unaware if they were in the experimental or control condition, similar to using a taste-matching agent in a drug trial
Who Masked: Participant
Masking Description: The participants will be unaware of what group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Active Comparator): There will be six, one hour, treatment sessions across nine weeks of a mindfulness intervention program, a post treatment assessment, and a follow up assessment three months later. The sessions will occur over zoom with a trained member of the study staff.
  Interventions: Behavioral: Mindfulness
- EmRes (Experimental): There will be six, one hour, treatment sessions across nine weeks of an Emotional Resolution therapy intervention program, a post treatment assessment, and a follow up assessment three months later. The sessions will occur over zoom with a trained emotional resolution coach.
  Interventions: Behavioral: EmRes

INTERVENTIONS:
Behavioral: EmRes — There will be six, one hour, treatment sessions across nine weeks of emotional resolution therapy, a post treatment assessment, and a follow up assessment three months later. The sessions will occur over zoom with a licensed therapist.
  Arms: EmRes
Behavioral: Mindfulness — There will be six, one hour, treatment sessions across nine weeks of a mindfulness intervention program, a post treatment assessment, and a follow up assessment three months later. The sessions will occur over zoom with a trained member of the study staff.
  Arms: Mindfulness

SUMMARY:
The purpose of the study is to conduct an initial test of the efficacy of Emotional Resolution (EmRes) therapy to reduce anxiety in healthcare workers. The investigators hypothesize EmRes will reduce levels of anxiety in participants compared to an active control group engaged in mindfulness-based gratitude.

DETAILED DESCRIPTION:
More than 1 in 5 adults in the US live with a mental illness, however, treatment is inaccessible to many. In fact, 63% of Californians with a mental health disorder do not receive treatment. Those who do receive treatment are burdened with long wait times. For example, the National Council of Mental Wellbeing reports the average wait time to access behavioral health services is currently about six weeks. Health care workers have been particularly affected by the inaccessibility of mental health treatment options, with nearly half of healthcare workers experiencing burnout during the COVID-19 pandemic. Therefore it is important to explore new types of effective and accessible therapeutic techniques.

Many different therapeutic techniques are emerging that may expand the toolkit of mental healthcare providers to allow them to deliver new solutions to their patients. For example, therapeutic programs which target emotion regulation have been found to increase the efficacy of more traditional psychotherapy. Here, the investigators seek to test the efficacy of one such therapeutic technique, Emotional Resolution therapy, at reducing anxiety in healthcare workers. Because this therapeutic technique is delivered via zoom, and typically consists of only 6-8 sessions, it offers a promising solution to those seeking treatment in a more accessible and less burdensome way. If effective at reducing anxiety in healthcare workers, this therapeutic technique may reduce the burden on mental healthcare providers and help deal with the mental health crisis that is causing healthcare workers to quit due to burnout and burdening our society.

The investigators will recruit healthcare workers with anxiety to participate in the study who will be randomly assigned to complete either the target therapeutic or control intervention. Participants will be asked to participate in a baseline assessment and six one-hour treatment sessions across 9 weeks, a post treatment assessment, and a follow up assessment three months later. The investigators will collect micro blood samples and will provide a smart watch as compensation for their participation, which they will ask participants to wear throughout the duration of the study. Participants do not need to come into the lab to participate. All research activities will occur online, and devices and samples will be mailed.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to provide written informed consent
2. > 18 years of age at Visit
3. Fluent in English
4. Current healthcare worker in a hospital
5. Generalized anxiety disorder (GAD) score of > 5

Exclusion Criteria:

1. Unable to provide written informed consent
2. Under the age of 18
3. Not fluent in English
4. Not working as a healthcare worker in a hospital
5. GAD score < 5
6. Currently on anxiety medication (Beta Blockers or Benzodiazepines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
EmRes Efficacy - anxiety change at follow-up 1 | Baseline to Follow-up 1 (9 weeks)
  The purpose of the study is to conduct an initial test of the efficacy of EmRes therapy to change anxiety levels in healthcare workers. The investigators hypothesize EmRes will change levels of anxiety from baseline to follow-up 1 in participants compared to an active control group engaged in mindfulness-based gratitude. This will be measured by the 8 item PROMIS Anxiety Short form. Responses to each item are summed. Scores range from 8-40, with a higher score indicating higher anxiety. A statistically significant decrease from baseline to follow-up one in anxiety scores is a positive outcome.
EmRes Efficacy - anxiety change at follow-up 2 | Baseline to Follow-up 2 (18 weeks)
  The purpose of the study is to conduct an initial test of the efficacy of EmRes therapy to change in healthcare workers. The investigators hypothesize EmRes will change levels of anxiety from baseline to follow-up 2 in participants compared to an active control group engaged in mindfulness-based gratitude. This will be measured by the 8 item PROMIS Anxiety Short form. Responses to each item are summed. Scores range from 8-40, with a higher score indicating higher anxiety. A statistically significant decrease from baseline to follow-up two in anxiety scores is a positive outcome.

SECONDARY OUTCOMES:
Perceived stress change at follow-up 1 | Baseline to Follow-up 1 (9 weeks)
  The Perceived Stress Scale (PSS) is used to measure the perception of stress. That is, the degree to which situations in one's life are appraised as stressful.
  PSS scores are computed by summing ten items. Items 4, 5, 7, and 8 are reverse-scored. The range of the PSS-10 is 0-40, with higher scores indicating more perceived stress. As such, a statistically significant decrease in PSS-10 scores from baseline to follow-up one indicates decreased stress and is a positive outcome.
Perceived stress change at follow-up 2 | Baseline to Follow-up 2 (18 weeks)
  The Perceived Stress Scale (PSS) is used to measure the perception of stress. That is, the degree to which situations in one's life are appraised as stressful.
  PSS scores are computed by summing ten items. Items 4, 5, 7, and 8 are reverse-scored. The range of the PSS-10 is 0-40, with higher scores indicating more perceived stress. As such, a statistically significant decrease in PSS-10 scores from baseline to follow-up two indicates decreased stress and is a positive outcome.
Burnout change at follow-up 1 | Baseline to Follow-up 1 (9 weeks)
  Burnout will be measured by The Maslach Burnout Inventory (MBI) which contains 22 symptom items pertaining to occupational burnout. Investigators will sum the first two sections (where higher scores represent a negative outcome) and balance this against the third section (where higher scores represent a positive outcome). Scores will be calculated as a ratio: Exhaustion+Depersonalization:Personal Achievement. High ratios reflect more burnout, and low ratios reflect less burnout. A statistically significant reduction in burnout from baseline to follow-up 1 represents a positive outcome.
  Exhaustion: 6 items, scores are summed, with a range of 0-36 possible. Higher scores = more exhaustion/burnout Depersonalization: 7 items, scores are summed, with a range of 0-42 possible. Higher scores = more depersonalization/burnout Personal achievement: 8 items, scores are summed, with a range of 0-48 possible. Higher scores = more personal achievement/less burnout
Burnout change at follow-up 2 | Baseline to Follow-up 2 (18 weeks)
  Burnout will be measured by The Maslach Burnout Inventory (MBI) which contains 22 symptom items pertaining to occupational burnout. Investigators will sum the first two sections (where higher scores represent a negative outcome) and balance this against the third section (where higher scores represent a positive outcome) . Scores will be calculated as a ratio: Exhaustion+Depersonalization:Personal Achievement. High ratios reflect more burnout, and low ratios reflect less burnout. A statistically significant reduction in burnout from baseline to follow-up 2 represents a positive outcome.
  Exhaustion: 6 items, scores are summed, with a range of 0-36 possible. Higher scores = more exhaustion/burnout Depersonalization: 7 items, scores are summed, with a range of 0-42 possible. Higher scores = more depersonalization/burnout Personal achievement: eight items, scores are summed, with a range of 0-48 possible. Higher scores = more personal achievement/less burnout

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Berking M, Wupperman P, Reichardt A, Pejic T, Dippel A, Znoj H. Emotion-regulation skills as a treatment target in psychotherapy. Behav Res Ther. 2008 Nov;46(11):1230-7. doi: 10.1016/j.brat.2008.08.005. Epub 2008 Aug 30. PMID 18835479
- [Background] Schnell K, Herpertz SC. Emotion Regulation and Social Cognition as Functional Targets of Mechanism-Based Psychotherapy in Major Depression With Comorbid Personality Pathology. J Pers Disord. 2018 Jan;32(Suppl):12-35. doi: 10.1521/pedi.2018.32.supp.12. PMID 29388896
- [Background] Ghahramani S, Lankarani KB, Yousefi M, Heydari K, Shahabi S, Azmand S. A Systematic Review and Meta-Analysis of Burnout Among Healthcare Workers During COVID-19. Front Psychiatry. 2021 Nov 10;12:758849. doi: 10.3389/fpsyt.2021.758849. eCollection 2021. PMID 34858231
- [Background] Fresco DM, Mennin DS, Heimberg RG, Ritter M. Emotion Regulation Therapy for Generalized Anxiety Disorder. Cogn Behav Pract. 2013 Aug;20(3):282-300. doi: 10.1016/j.cbpra.2013.02.001. PMID 27499606
- See also: California Health Care Foundation — https://www.chcf.org/